CLINICAL TRIAL: NCT00682110
Title: Comparing Different Methods For Measurement of Cardiac Output During Orthotopic Liver Transplantation
Brief Title: Hemodynamic Measurements During Liver Transplantation
Acronym: OLT
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Ivan Kangrga, MD, PhD, Professor of Anesthesiology
Other Study IDs: 07-0042
Record Dates: First submitted 2008-05-16; First posted 2008-05-22 (Estimated); Last update posted 2010-04-01 (Estimated); Status verified 2010-03

CONDITIONS: Liver Transplantation
Keywords: End-stage liver disease; Hemodynamic measurements; Hyperdynamic circulation; Pulmonary artery catheter; Cardiac output
MeSH Terms: conditions — End Stage Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to determine if the less invasive monitors are as reliable for measuring heart function in patients undergoing liver transplantation as the more invasive pulmonary artery.

DETAILED DESCRIPTION:
Pulmonary artery catheter (PAC)is considered the gold standard in monitoring of heart function during orthotopic liver transplantation (OLT). Placement of PAC is very invasive (it passes thorough the heart chambers and into the pulmonary artery) and its benefits on the outcomes have not been proven. This study compares two newer FDA approved much less invasive devices to the PAC. The two new devices assess the heart function based either on the peripheral arterial waveform alone (Vigileo, Edwards Lifesciences)or the combination of peripheral arterial waveform and chemical indicator dilution (LiDCO, Cambridge, UK).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Scheduled for liver transplantation
* Patient undergoing vascular surgery where invasive arterial pressure is indicated (control subjects)

Exclusion Criteria:

* We will exclude patients taking lithium based medication
* Patients who weigh less than 40 kg; AND
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 subjects will be enrolled in this observational study in the Liver Transplant Group; 10 patients in the Other Surgery Control Group for a total of 30 subjects. Patients will be recruited from the Operating Room schedule. Written, informed consent will be obtained from each subject prior to surgery. All participants will be informed that they may decline to participate in, or withdraw from, the study at any time.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-07; Primary Completion 2009-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Agreement between cardiac output measurements obtained with PAC, Vigileo and LiDCO | Specific phases of liver transplantation surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Kangrga, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Vannucci A, Burykin A, Krejci V, Peck T, Buchman TG, Kangrga IM. Postreperfusion cardiac arrest and resuscitation during orthotopic liver transplantation: dynamic visualization and analysis of physiologic recordings. Shock. 2012 Jan;37(1):34-8. doi: 10.1097/SHK.0b013e318239b128. PMID 22089184
- [Derived] Krejci V, Vannucci A, Abbas A, Chapman W, Kangrga IM. Comparison of calibrated and uncalibrated arterial pressure-based cardiac output monitors during orthotopic liver transplantation. Liver Transpl. 2010 Jun;16(6):773-82. doi: 10.1002/lt.22056. PMID 20517912
- [Derived] Vannucci A, Krejci V, Kangrga I. Performance of Vigileo and LiDCOplus cardiac output monitors during a prolonged cardiac arrest and resuscitation. Eur J Anaesthesiol. 2009 Oct;26(10):885-7. doi: 10.1097/EJA.0b013e32832fa5db. No abstract available. PMID 19606043